CLINICAL TRIAL: NCT04565327
Title: Hyperpolarized 13C Pyruvate MRI for Treatment Response Assessment in Pancreatic Ductal Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Zhen Wang, MD (Other)
Responsible Party: Sponsor-Investigator, Zhen Wang, MD, Professor in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20925; NCI-2020-06080 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Hyperpolarized 13C Pyruvate; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Single Dose/Image (Experimental): Patients receive hyperpolarized carbon C 13 pyruvate intravenously (IV) over less than one minute then undergo MRI over 5 minutes at baseline
  Interventions: Drug: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Imaging (MRI)
- Cohort B: Multiple Dose/Images (Experimental): Patients receive hyperpolarized carbon C 13 pyruvate IV over less than one minute then undergo MRI over 5 minutes at baseline and 4 weeks after beginning treatment
  Interventions: Drug: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Drug: Hyperpolarized Carbon C 13 Pyruvate — Given IV prior to imaging
  Other Names: Hyperpolarized 13C Pyruvate
Procedure: Magnetic Resonance Imaging (MRI) — Undergo MRI
  Other Names: MRI; Magnetic Resonance Imaging Scan; MR Imaging

SUMMARY:
This phase II trial investigates whether magnetic resonance imaging (MRI) using hyperpolarized carbon-13 (13C) pyruvate can be useful for evaluating early treatment response in patients with pancreatic cancer that has spread to nearby tissue or lymph nodes (locally advanced) or spread to other places in the body (metastatic). Hyperpolarized 13C pyruvate is different from standard clinical MRI contrast (e.g. gadolinium) in that it provides information on how a tumor processes nutrients. MRI is used to see tumor uptake and breakdown of hyperpolarized carbon-13 pyruvate molecules, which can tell how the tumor processes nutrients. Hyperpolarized 13C pyruvate MRI may help in understanding how the tumor responds to the treatments patients may be receiving.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the signal-to-noise ratio of 13C pyruvate metabolism (peak 13C lactate/pyruvate ratio, 13C lactate/pyruvate area-under-the-curve (AUC) ratio, and apparent rate constant for pyruvate-to-lactate conversion, kPL) in the target tumor (primary tumor and/or abdominal metastases) in Cohort A.

II. To determine the percent changes in the target tumor (primary tumor and/or abdominal metastases) 13C pyruvate metabolism (peak 13C lactate/pyruvate ratio, 13C lactate/pyruvate AUC ratio, and kPL) between pre-treatment scan and scan obtained at 4-week (+/-2 weeks) following treatment initiation in Cohort B.

SECONDARY OBJECTIVES:

I. To determine the repeatability of 13C pyruvate metabolism measures in the target tumor (primary tumor and/or abdominal metastasis) in patients with same-day repeated dose in Cohort A and B.

II. To determine whether the baseline or the changes in the target tumor (primary tumor and/or abdominal metastases) 13C pyruvate metabolism at 4 weeks following treatment initiation are associated with the best objective response as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria on subsequent clinical computed tomography (CT) scans in Cohort B.

EXPLORATORY OBJECTIVE:

I. To explore 13C pyruvate metabolism between the primary tumor and abdominal metastases (when present) both at baseline and following treatment in both Cohort A and B.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients receive hyperpolarized carbon C 13 pyruvate intravenously (IV) over less than one minute then undergo MRI over 5 minutes at baseline in the absence of unacceptable toxicity.

COHORT B: Patients receive hyperpolarized carbon C 13 pyruvate IV over less than one minute then undergo MRI over 5 minutes at baseline and 4 weeks after beginning treatment in the absence of unacceptable toxicity.

In both cohorts, patients may receive an optional second hyperpolarized carbon C 13 pyruvate dose and undergo MRI within 15 to 60 minutes following the completion of the first scan.

After completion of study treatment, patients are followed up every 2-3 months

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic pancreatic ductal adenocarcinoma, with at least one target lesion in the abdomen measuring >= 1 cm
* The subject is able and willing to comply with study procedures and provide signed and dated informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Patients who because of age, general medical or psychiatric condition, or physiologic status cannot give valid informed consent
* Patients unwilling or unable to undergo magnetic resonance (MR) imaging, including patients with contraindications to MRI, such as cardiac pacemakers or non-compatible intracranial vascular clips
* Poorly controlled hypertension, defined as either systolic > 170 or diastolic > 110. The addition of anti-hypertensives to control blood pressure is allowed for eligibility determination
* Congestive heart failure >= class III
* Myocardial infarction within the past year
* History of QT prolongation on electrocardiogram (EKG), defined as pretreatment QTs > 440 msec in males or > 460 msec in females
* Pregnant and lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gordon JW, Chen HY, Nickles T, Lee PM, Bok R, Ohliger MA, Okamoto K, Ko AH, Larson PEZ, Wang ZJ. Hyperpolarized 13C Metabolic MRI of Patients with Pancreatic Ductal Adenocarcinoma. J Magn Reson Imaging. 2024 Aug;60(2):741-749. doi: 10.1002/jmri.29162. Epub 2023 Dec 2. PMID 38041836

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were assigned to Cohort A based on diagnosis
Groups:
- Cohort A: Single Dose/Image: Participants receive hyperpolarized carbon C 13 pyruvate intravenously (IV) over less than one minute then undergo MRI over 5 minutes at baseline
- Cohort B: Multiple Dose/Images: Participants receive hyperpolarized carbon C 13 pyruvate IV over less than one minute then undergo MRI over 5 minutes at baseline and 4 weeks after beginning treatment
Period: Overall Study
Arm/Group | Cohort A: Single Dose/Image | Cohort B: Multiple Dose/Images
Started | 0 | 7
Completed | 0 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were assigned to Cohort A
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Single Dose/Image | Cohort B: Multiple Dose/Images | Total
Number analyzed (Participants) | 0 | 7 | 7
Age, Customized [Count of Participants; unit: Participants]
  50-59 years old | 0 | 2 | 2
  60-69 years old | 0 | 4 | 4
  70-79 years old | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 0 | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 0 | 6 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 3 | 3
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States |  | 7 | 7

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Signal-to-noise Ratio of the Target Lesion 13C Pyruvate Metabolism Measures Will be Determined for Each Patient
Description: Descriptive statistics will be used to summarize the mean, standard deviation, and 95% confidence interval of the measurements.
Time Frame: Baseline
Population: No participants were enrolled to Cohort A
Arm/Group | Cohort A: Single Dose/Image
Number analyzed (Participants) | 0

2. Primary Outcome: Cohort B: Target Tumor Metabolism
Description: Paired t-test or Wilcoxon signed rank test will be used to compare the target tumor Hyperpolarized (HP) 13C pyruvate metabolism pre- and 4-week (+/- 2 weeks) post treatment initiation.
Time Frame: Up to 4 weeks
Population: Data was not collected for this endpoint
Arm/Group | Cohort B: Multiple Dose/Images
Number analyzed (Participants) | 0

3. Secondary Outcome: Cohort A: Intraclass Correlation Coefficient (ICC)
Description: ICC will be used to estimate the intra-subject agreement to assess repeatability of tumor HP 13C pyruvate metabolism in patients with same-day repeated dose. ICC will also be used to estimate agreement obtained from a one-way analysis of variance model based on 2 measurements per subject. The result will be presented with a 95% confidence interval
Time Frame: Up to 6 months
Population: No participants were enrolled to Cohort A
Arm/Group | Cohort A: Single Dose/Image
Number analyzed (Participants) | 0

4. Secondary Outcome: Cohort B: Best Objective Response
Description: Objective response for patients in Cohort B will be defined using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 on subsequent clinical CT scans. For the purpose of response assessment in this pilot study, we will group patients either as having disease control when the best response is complete response (CR), partial response (PR), or stable disease (SD) on subsequent clinical CT scans, or having disease progression when the best response is progressive disease (PD) on subsequent CT scans. Comparisons the baseline or changes in the target tumor 13C pyruvate metabolism at 4 weeks (+/-2 weeks) after treatment initiation between the disease control group and disease progression group (as defined by RECIST on subsequent clinical CT scans) will be made using the Mann-Whitney tests.
Time Frame: Up to 4 weeks after treatment initiation
Population: Data was not collected for this endpoint
Arm/Group | Cohort B: Multiple Dose/Images
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Description: No participants were enrolled under Cohort A
Arm/Group | Cohort A: Single Dose/Image | Cohort B: Multiple Dose/Images
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/7
Other Adverse Events (participants affected / at risk) | 0/0 | 0/7

LIMITATIONS AND CAVEATS:
Study closed earlier than expected due to slow accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT04565327/Prot_SAP_000.pdf